CLINICAL TRIAL: NCT00262301
Title: A Randomized, Placebo-controlled, Double-blind Phase III Study of the Efficacy and Safety of Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Brief Title: Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1 1304-01
Record Dates: First submitted 2005-12-01; First posted 2005-12-06 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Hereditary Angioedema; Angioneurotic Edema; Genetic Disorders
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Genetic Diseases, Inborn | interventions — Complement C1 Inhibitor Protein; conestat alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 IU/kg "rhC1INH" (Experimental): 100 IU/kg recombinant human C1 inhibitor
  Interventions: Drug: recombinant human C1 inhibitor
- Saline (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human C1 inhibitor — IV
  Other Names: "rhC1INH"; Ruconest; conestat alfa
  Arms: 100 IU/kg "rhC1INH"
Drug: Placebo — IV
  Other Names: saline; physiological salt solution
  Arms: Saline

SUMMARY:
Hereditary angioedema ("HAE") is a genetic disorder characterized by sudden recurrent attacks of local swelling (angioedema). These attacks are often painful and disabling, and, in some cases, life-threatening. "HAE" is caused by mutations in the "C1INH" gene that leads to a decrease in the blood level of functional "C1INH". This multi-center study was designed to assess the safety and tolerability, efficacy and pharmacodynamics/ pharmacokinetics of recombinant human C1 inhibitor ("rhC1INH") in the treatment of acute hereditary angioedema attacks.

DETAILED DESCRIPTION:
A prospectively planned interim analysis will be performed on the double-blind data.

ELIGIBILITY:
Inclusion Criteria:

* Clear clinical and laboratory diagnosis of HAE
* Baseline plasma level of functional C1INH of less than 50% of normal
* Evidence for exacerbation or development of a severe abdominal, oro-facial/ pharyngeal/ laryngeal, genito-urinary and/or peripheral HAE attack

Exclusion Criteria:

* Acquired angioedema
* Pregnancy or breastfeeding
* Participation in another clinical study within prior 3 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-06; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nuijens, MD, PhD, Study Chair — Pharming Group N.V.
Locations (2):
- For information on sites, please contact Pharming Medical Affairs Deparment, Leiden, Netherlands
- Emergency County Hospital, Internal Medicin Clinica, Allergology-Immunology Department, Târgu Mureş, Romania

REFERENCES:
- [Result] Zuraw B, Cicardi M, Levy RJ, Nuijens JH, Relan A, Visscher S, Haase G, Kaufman L, Hack CE. Recombinant human C1-inhibitor for the treatment of acute angioedema attacks in patients with hereditary angioedema. J Allergy Clin Immunol. 2010 Oct;126(4):821-827.e14. doi: 10.1016/j.jaci.2010.07.021. PMID 20920772
- [Result] Moldovan D, Reshef A, Fabiani J, Kivity S, Toubi E, Shlesinger M, Triggiani M, Montinaro V, Cillari E, Realdi G, Cancian M, Visscher S, Zanichelli A, Relan A, Cicardi M. Efficacy and safety of recombinant human C1-inhibitor for the treatment of attacks of hereditary angioedema: European open-label extension study. Clin Exp Allergy. 2012 Jun;42(6):929-35. doi: 10.1111/j.1365-2222.2012.03984.x. PMID 22909164
- [Derived] Bernstein JA, Relan A, Harper JR, Riedl M. Sustained response of recombinant human C1 esterase inhibitor for acute treatment of hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2017 Apr;118(4):452-455. doi: 10.1016/j.anai.2017.01.029. Epub 2017 Mar 9. PMID 28284978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the double-blind phase of the study, patients were randomized once to receive 100 IU/kg "rhC1INH" or Saline in a ratio of 1:1. After conclusion of the double-blind phase, patients with subsequent eligible attacks could be treated with open-label 1 vial (2100 IU) of "rhC1INH".
Pre-assignment Details: Patients could be enrolled into the open-label phase of the study after conclusion of the double-blind phase.
Groups:
- 100 IU/kg "rhC1INH": Includes all subjects randomized and who received 100 IU/kg recombinant human C1 inhibitor in the double-blind phase.
- Saline: Includes all subjects randomized and who received Saline solution in the double-blind phase.
- 1 Vial (2100 IU) "rhC1INH": Includes all subjects who received, 1 vial (2100 IU) open-label "rhC1INH" in the open-label extension phase. Patients received 1 vial initially and could receive an additional 1-2 vials within 4 hours at the investigator's discretion.
Period: Double-blind Phase
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH"
Started | 16 | 16 | 0
Completed | 15 | 15 | 0
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — worsening of "HAE" symptoms | 0 | 1 | 0
Period: Open-label Phase
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH"
Started | 0 | 0 | 57 (14/57 patients crossed over from the double-blind phase (7/14 were treated with 100 U/kg "rhC1INH"))
Completed | 0 | 0 | 57
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 100 IU/kg "rhC1INH": Includes all subjects randomized who received 100 IU/kg recombinant human C1 inhibitor in the double-blind phase.
- 1 Vial (2100 IU) "rhC1INH": Includes all subjects who received 1 vial (2100 IU) open-label "rhC1INH" in the open-label extension phase.
- Total: Total of all reporting groups
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH" | Total
Number analyzed (Participants) | 16 | 16 | 43 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 9 | 11
  Between 18 and 65 years | 13 | 12 | 33 | 58
  >=65 years | 2 | 3 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 28 | 45
  Male | 8 | 7 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Relief of Symptoms
Description: The time to beginning of relief of symptoms has been assessed by using a patient-reported visual analogue scale ("VAS") ranging from 0 mm (no symptoms at all) to 100 mm (extremely disabling). Time to beginning of relief of symptoms at the location that showed first "VAS" score decrease of at least 20 mm from baseline score (t= 0 min) to the next assessment time-point). Assessment time-points were taken on pre-scheduled time-points after drug administration: baseline (0 minutes), 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 48 hours. Time to beginning of relief has been calculated as median time, by using the exact time-points on which each assessment was performed.
Time Frame: up to 48 hours after study drug administration
Population: The full analysis set ("FAS" or "mITT") was defined as the set of patients who provided Informed Consent, were randomized and took at least one dose of the study drug administration.
Measure: Median (Full Range); unit: minutes
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH"
Number analyzed (Participants) | 16 | 16 | 57
minutes | 62 [15 to 1470] | 508 [15 to 2880] | 61 [15 to 1455]
Statistical Analysis 1: Comparison: 100 IU/kg "rhC1INH" vs Saline; Test type: Superiority or Other; p = 0.003, Log Rank

2. Secondary Outcome: Time to Minimal Symptoms
Description: the time to minimal symptoms was the time to minimal symptoms for an attack, assessed using the Visual Analogue Scale ("VAS") score. Symptoms were said to be minimal when the "VAS" score at all locations was below 20 mm. Assessment time-points were: baseline (0 minutes), 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours, 48 hours. Time to minimal symptoms has been calculated by using the exact time-points on which each assessment was performed.
Time Frame: up to 48 hours after study drug administration
Population: The full analysis set ("FAS" or "mITT") was defined as the set of patients who provided Informed Consent, were randomized and took at least one dose of study drug administration.
Measure: Median (Full Range); unit: minutes
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH"
Number analyzed (Participants) | 16 | 16 | 57
minutes | 480 [15 to 2400] | 1440 [31 to 2885] | 241 [15 to 4333]
Statistical Analysis 1: Comparison: 100 IU/kg "rhC1INH" vs Saline; Test type: Superiority or Other; p = 0.005, Log Rank

ADVERSE EVENTS:
Time Frame: Treatment-Emergent-Adverse-Events ("TEAEs") were defined as events with start from onset of study drug administration. Serious Adverse events and Adverse events for each arm with onset dates within 7 days of study drug administration have been listed.
Arm/Group | 100 IU/kg "rhC1INH" | Saline | 1 Vial (2100 IU) "rhC1INH"
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/16 | 0/57
Other Adverse Events (participants affected / at risk) | 2/16 | 5/16 | 6/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 IU/kg "rhC1INH" (N=16) | Saline (N=16) | 1 Vial (2100 IU) "rhC1INH" (N=57)
Prostate examination (Investigations) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 IU/kg "rhC1INH" (N=16) | Saline (N=16) | 1 Vial (2100 IU) "rhC1INH" (N=57)
headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
pain (General disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to its submission or disclosure. The sponsor may request to delete information identified by sponsor as confidential information prior to submitting such manuscript and/or abstract for publication. For a multi-center study, the investigator must wait (i) at least 24 months after the study is completed at all sites or (ii) until after the multi-center publication.